CLINICAL TRIAL: NCT00424775
Title: A Phase I Study of Carboplatin + Paclitaxel and MK0683 in Patients With Chemotherapy-naive Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Carboplatin + Paclitaxel and MK0683 in Patients With Chemotherapy-naive Non-Small Cell Lung Cancer (NSCLC)(0683-066)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0683-066; 2007_001
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Results first posted 2009-06-01 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-03

CONDITIONS: Neoplasms
Keywords: Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Vorinostat

INTERVENTIONS:
Drug: MK0683, vorinostat — vorinostat 300 mg or 400 mg once daily consecutive days (14 days) followed by 11 days of rest in the first cycle or 7 days of rest in the second or later cycle.
  Other Names: MK0683

SUMMARY:
The clinical study will evaluate safety, tolerability and Pharmacokinetics of MK0683 in combination with carboplatin and paclitaxel in chemotherapy-naive NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* Chemotherapy-naive patients who are histologically or cytologically diagnosed NSCLC with stage IIIB (not applicable of radical thoracic radiation) or stage IV
* Patients with normal organ function and bone marrow function

Exclusion Criteria:

* Given radical thoracic radiation for NSCLC or radiation for other than original lesion within 3 weeks
* Any peripheral neuropathy above grade 2
* Any ascites, pleural effusion or pericardiac effusion which requires treatment
* Any uncontrolled concomitant illness
* Pregnant or breast-feeding

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first participant in: 26 January 2007. Data of last participant's last visit in study protocol: 7 March 2007. The study was conducted at single center in Japan.
Pre-assignment Details: Vorinostat with Carboplatin and Paclitaxel were investigated in participants with chemotherapy-naive non-small cell lung cancer.
  Enroll 3 participants to dose level 1 of vorinostat and decide whether to enroll additional participants based on the Dose Limited Toxicity (DLT) manifestation.
  The starting dose of vorinostat was 300 mg once daily.
Groups:
- Vorinostat (300 mg): This group includes data from all participants who were treated with vorinostat 300 mg once daily consecutive days (14 days) followed by 11 days of rest in the first cycle or 7 days of rest in the second or later cycle.
- Vorinostat (400 mg): This group includes data from all participants who are treated with vorinostat 400 mg once daily consecutive days (14 days) followed by 11 days of rest in the first cycle or 7 days of rest in the second or later cycle. However, no participants received vorinostat 400 mg once daily due to early discontinuation of the study based on the dose limited toxicity on vorinostat 300 mg once daily.
Period: Overall Study
Arm/Group | Vorinostat (300 mg) | Vorinostat (400 mg)
Started | 3 | 0
Completed | 0 | 0
Not Completed | 3 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Vorinostat (300 mg): This group includes data from all participants who were treated with vorinostat 300 mg once daily consecutive days (14 days) followed by 11 days of rest (first cycle).
Arm/Group | Vorinostat (300 mg)
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Dose Limited Toxicity at First Cycle
Description: Dose Limited Toxicity = Drug-related side effects that are serious enough to prevent an increase in dose or level of that treatment.
Time Frame: 25 Days (first cycle)
Population: All participants who received vorinostat 300 mg once daily.
Measure: Number; unit: Participants
Arm/Group | Vorinostat (300 mg)
Number analyzed (Participants) | 3
Participants | 3

2. Secondary Outcome: Area Under the Curve (AUC(0-24 hr)) at Day 4
Description: Area Under the Curve (AUC (0-24 hr)) = Area under the plasma concentration versus time curve (AUC) from time zero to 24 hour.
Time Frame: Day 4
Population: Participants who received vorinostat 300 mg once daily and had Pharmacokinetics Data on Day 4.
Measure: Mean (Full Range); unit: µM hr
Arm/Group | Vorinostat (300 mg)
Number analyzed (Participants) | 2
µM hr | 9.76 [6.61 to 12.90]

3. Secondary Outcome: Area Under the Curve (AUC(0-24 hr)) at Day 5
Description: as for outcome 2
Time Frame: Day 5
Population: Participants who received vorinostat 300 mg once daily and had Pharmacokinetics Data on Day 5.
Measure: Mean (Full Range); unit: µM hr
Arm/Group | Vorinostat (300 mg)
Number analyzed (Participants) | 2
µM hr | 6.26 [5.37 to 7.14]

4. Secondary Outcome: Maximum Concentration (Cmax) at Day 4
Description: Maximum Concentration (Cmax) = the maximum plasma concentration of the drug
Time Frame: Day 4
Population: Participants who received vorinostat 300 mg once daily and had Pharmacokinetics Data on Day 4.
Measure: Mean (Full Range); unit: µM
Arm/Group | Vorinostat (300 mg)
Number analyzed (Participants) | 2
µM | 1.54 [0.99 to 2.09]

5. Secondary Outcome: Maximum Concentration (Cmax) at Day 5
Description: Maximum Concentration (Cmax) = the maximum plasma concentration of the drug
Time Frame: Day 5
Population: Participants who received vorinostat 300 mg once daily and had Pharmacokinetics Data on Day 5.
Measure: Mean (Full Range); unit: µM
Arm/Group | Vorinostat (300 mg)
Number analyzed (Participants) | 2
µM | 1.96 [1.60 to 2.32]

ADVERSE EVENTS:
Arm/Group | Vorinostat (300 mg)
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Vorinostat (300 mg)
Anaemia (Blood and lymphatic system disorders) | 2/3
Leukopenia (Blood and lymphatic system disorders) | 2/3
Lymphopenia (Blood and lymphatic system disorders) | 2/3
Diarrhoea (Gastrointestinal disorders) | 2/3
Nausea (Gastrointestinal disorders) | 2/3
Vomiting (Gastrointestinal disorders) | 2/3
Fatigue (General disorders) | 2/3
Pyrexia (General disorders) | 2/3
Anorexia (Metabolism and nutrition disorders) | 2/3
Neutrophil count decreased (Investigations) | 2/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.